CLINICAL TRIAL: NCT02983903
Title: An Un-blinded, Intra-patient Comparison of Transbronchial Forceps Biopsy and Cryobiopsy for Peripheral Pulmonary Lesions
Brief Title: Cryobiopsy Versus Forceps Biopsy for Pulmonary Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis also showed a lack of benefit in the experimental arm.
Sponsor: University of Pennsylvania (Other)
Collaborators: Andrew Haas (Unknown); Anil Vachani (Unknown); Anthony Lanfranco (Unknown); Kevin Ma (Unknown); Jeffrey Thompson (Unknown); Edmund Moon (Unknown)
Responsible Party: Principal Investigator, David DiBardino, Assistant Professor of Clinical Medicine, Section of Interventional Pulmonology and Thoracic Oncology, Assistant Professor of Medicine at the Hospital of the University of Pennsylvania, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB # 825506
Record Dates: First submitted 2016-11-21; First posted 2016-12-06 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single intervention arm - transbronchial biopsy (Experimental): Patients enrolled in this single arm study will have lung nodules biopsied by traditional forceps followed by transbronchial cryobiopsy
  Interventions: Procedure: transbronchial biopsy

INTERVENTIONS:
Procedure: transbronchial biopsy

SUMMARY:
Purpose: Patients with peripheral lung nodules require evaluation for lung cancer. Our aim is to assess the diagnostic yield of a new technique, transbronchial cryobiopsies, in patients at risk for lung cancer. Target population: Patients referred for bronchoscopy and lung biopsies as a part of their work up for peripheral lung lesions. Procedures: Patients enrolled will have forceps transbronchial biopsies followed by transbronchial cryobiopsies for their lung lesion during bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18
2. At least one peripheral lung lesion >8mm documented on CT scan referred for diagnostic bronchoscopy
3. Subject is able to undergo informed consent

Exclusion Criteria:

1. Coagulopathy (platelet count < 50,000, INR > 1.5) detected on blood testing done within 6 weeks of the procedural visit
2. Lesion associated with a prominent vessel evident on CT scan
3. Pure ground glass lesion
4. Fibrotic interstitial lung abnormalities on chest CT
5. Bullous emphysema in region of nodule
6. Supplemental oxygen utilization at baseline
7. BMI > 40
8. End stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
The increase in sensitivity for diagnosing lung cancer with the addition of cryobiopsy to standard forceps biopsy for a suspicious lung nodule. | 1 year
  Sensitivity for cancer is defined as true positives / (true positives + false negatives) with respect to diagnosing malignancy. If the bronchoscopic procedure fails to diagnose malignancy, the gold standard will be the results of any further, more invasive testing that is clinically indicated to evaluate the nodule.

SECONDARY OUTCOMES:
The increase in sensitivity for diagnosing a specific benign lung disease with the addition of cryobiopsy to standard forceps biopsy for a suspicious lung nodule. | 1 year
  Sensitivity is defined as true positives / (true positives + false negatives) with respect to diagnosing a specific benign condition that is thought to represent the lung nodule seen on CT scan. If the bronchoscopic procedure fails to diagnose a specific benign condition, the gold standard will be the results of any further, more invasive testing and stable follow-up imaging at 1 year.
The number of participants with pneumothorax or significant bleeding related to the addition of transbronchial cryobiopsy to standard forceps biopsy. | 1 year
  A chest X-ray and ultrasound will be done to check for pneumothorax after standard forceps biopsy and after the addition of transbronchial cryobiopsy. Bleeding will be measured with a standardized scale (grade 0 = traces of blood not requiring suctioning; grade 1 = bleeding requiring suction to clear; grade 2 = bleeding requiring wedging of the biopsied segment with the flexible bronchoscope and/or iced saline/epinephrine; grade 3 = bleeding requiring further intervention such as balloon occlusion or inflation of the bronchial blocker; grade 4 = bleeding resulting in airway obstruction and acute hypoxemic respiratory failure, cardiopulmonary instability, transfusion of packed RBCs, and/or admission to the ICU) both after forceps biopsy and again after transbronchial cryobiopsy.

CONTACTS AND LOCATIONS:
Overall Officials: David M DiBardino, MD, Principal Investigator — University of Pennslyvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No